CLINICAL TRIAL: NCT05409001
Title: Falls From Sitting to Standing
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0850 SIUHN
Record Dates: First submitted 2022-05-23; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Falls, Tomography of the Head, Cervical Spine, Chest, Abdomen, and Pelvis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: tomography pan scan — This is a retrospective chart review

SUMMARY:
Background: When evaluating trauma patients, many centers perform computed tomography of the head, cervical spine, chest, abdomen, and pelvis, the so-called "pan-scan." Here, we evaluate the utility of pan-scan in geriatric patients who sustained ground-level falls.

Study Design: We performed a retrospective review of consecutive patients from the trauma registry of a large, urban Level 1 trauma center. Inclusion criteria were registration during the 2019 calendar year, age ≥ 65, mechanism of fall from either sitting or standing, and performance of "pan-scan" at time of assessment. Patient demographics, physical exam findings, CT results, injuries, and patient disposition were recorded. The sensitivity, specificity, positive and negative predictive values of the physical exam for significant injuries were calculated.

ELIGIBILITY:
Inclusion criteria

* age >65
* presented with fall from sitting or standing from 01/01/2019-12/31/2019

Exclusion criteria included

* age <65 years,
* falls from height,
* GCS less than 14,
* patients who did not undergo the complete pan-scan.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A retrospective chart review was conducted using the trauma registry at a large, urban Level 1 trauma center. This registry was queried for consecutive elderly patients (age >65 years) who presented with fall from sitting or standing from 01/01/2019-12/31/2019. This trauma registry includes all patients of which the trauma surgery team was notified as part of the insinuation's trauma notification protocol. It also includes patients who were ultimately admitted to the hospital with ICD 10 codes consistent with traumatic injuries, regardless of trauma team activation. Patients discharged from the Emergency Department with a traumatic injury may have limited data in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 751 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity of physical exam compared to CT scan and identifying traumatic injuries | 2 years
  Sensitivity of physical exam compared to CT scan and identifying traumatic injuries. Sensitivity is a statistical measure which was calculated using our SAS software as described in methods. CT scan was used as the gold standard. Both physical exam and CAT scan were performed on initial presentation with a time frame on the order of minutes to hours.
Prevalence of injury. | 2 years
  Traumatic injuries were determined by CT scan, tabulated, and broken down by body region as well as injury type. These data were collected at the time of CT scan on initial presentation. These data presented as whole numbers and percentages.
Disposition from ED | 2 years
  Dispositions were determined by chart review, tabulated, and broken down by disposition location. These data collected at the time of admission
Disposition from hospital. | 2 years
  Dispositions were determined by chart review, tabulated, and broken down by disposition location, including patient expiration in some cases. These data were collected at the time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- SIUH Northwell Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
aggregate data will be published